CLINICAL TRIAL: NCT04939220
Title: Supraglottic Airway Use for Transesophageal Echocardiography: a Safe Alternative to Deep Sedation for Patients With High-risk Cardiopulmonary Disease. (SGA-TEE)
Brief Title: SGA for TEE: Safe Alternative to Deep Sedation for Patients With High-risk Cardiopulmonary Disease.
Acronym: SGA-TEE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI unavailable to conduct study or begin recruitment. No longer feasible.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202101097
Record Dates: First submitted 2021-05-24; First posted 2021-06-25 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Cardiopulmonary Disease
Keywords: TEE; SGA; Anesthesia; sedation; Chronic Hypoxemic lung Disease; Obstructive Sleep Apnea; Morbid Obesity
MeSH Terms: conditions — Pulmonary Heart Disease; Sleep Apnea, Obstructive; Obesity, Morbid | interventions — Deep Sedation

STUDY DESIGN:
Intervention Model Description: Prospective, randomized control trial
Who Masked: Participant
Masking Description: Randomization to control group- deep sedation with propofol and natural airway or Experimental group-SGA Placement and maintenance with inhalational anesthetic or propofol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Deep sedation with propofol and natural airway
  Interventions: Procedure: TEE with Deep Sedation
- Experimental Group (Experimental): SGA Placement and maintenance with inhalational anesthetic or propofol
  Interventions: Procedure: TEE with SGA

INTERVENTIONS:
Procedure: TEE with SGA — SGA Placement and maintenance with inhalational anesthetic or propofol
  Arms: Experimental Group
Procedure: TEE with Deep Sedation — Deep sedation with propofol and natural airway
  Arms: Control Group

SUMMARY:
Increasingly, transesophageal echos (TEEs) are being done on high risk patients. A TEE is a short procedure done with deep sedation, but poses an increased risk of apnea/ hypoxemia in those with pulmonary disease. It is desirable to avoid intubation, which adds risk. Use of supraglottic airway (SGA) may offer an alternative. The investigators hypothesize that TEEs can be done successfully with an SGA in place. The investigators propose a prospective RCT to compare TEE exams done with deep sedation to those done with an SGA.

DETAILED DESCRIPTION:
Increasingly, non-operating room anesthesia (NORA) cases are being performed on patients with high risk for needing advanced airway management, ie patients with morbid obesity, chronic hypoxemic lung disease, obstructive sleep apnea.

Transesophageal echocardiography (TEE) exams are one example of this. While a TEE is typically a short, diagnostic procedure done with deep sedation, deep sedation poses an increased risk of hypoventilation and hypoxemia in patients with cardiopulmonary disease. It is desirable to avoid endotracheal intubation for TEE exams, as the procedure is short and can easily be done without muscle relaxation.

Moreover, securing the airway with an endotracheal tube (ETT) is not without significant risk. The use of a supraglottic airway (SGA) may offer an alternative for patients receiving a TEE who are high risk candidates for deep sedation with a natural airway.

The investigators hypothesize that the TEE procedure can be done successfully, without interruption, with an SGA in place. Our secondary hypothesis is that SGA use in high-risk patients may be safer than deep sedation, as there may be less episodes of hypoventilation and hypoxemia.

The investigators propose a prospective randomized control trial to compare TEE exams done with deep sedation (control group) to those done with SGA (intervention group). Our primary outcome will be TEE study completion, and secondary outcomes will focus on the safety profile of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults presenting for elective outpatient TEE examinations at UF Shands hospital during the study duration

Exclusion Criteria:

* Known or suspected difficult airway, patient refusal or inability to consent, patients to have emergent or urgent TEE exams, patients considered to have full stomach ie gastroparesis or achalasia

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-03-09 (Estimated); Study Completion 2024-03-09 (Estimated)

PRIMARY OUTCOMES:
The number of successfully completed TEE examinations with the assigned airway intervention | Duration of procedure
  The primary outcome is a binary data point (yes/no) defined as the success of using the assigned LMA or natural airway successfully for a TEE procedure.

SECONDARY OUTCOMES:
Ease of Placement of LMA | Duration of procedure
  Defined by placement of LMA on first attempt, with good chest rise on positive pressure assisted ventilation, no audible leak on assisted ventilation with cuff pressure <32 cm H2O, and sustained, square waveform capnography
Alternative Airway device | Duration of procedure
  this secondary outcome is a binary data point (yes/no) on the use of an endotracheal tube for rescue from failure of assigned airway type for the procedure (LMA vs natural airway with sedation)
Dislocation of LMA | Duration of procedure
  this secondary outcome is a binary data point (yes/no) for any form of dislocation of the LMA during the endoscopic procedure necessitating repositioning of the LMA.
Chin Lift or Jaw Thrust | Duration of Procedure
  this secondary outcome is a binary data point (yes/no) for the need to perform chin lift or jaw thrust to maintain a patent airway.
Pharyngeal Bleeding | Duration of Procedure
  the incidence of pharyngeal bleeding during placement or after the procedure
Hypoxia | Duration of Procedure
  Hypoxia during the procedure will be defined as an oxygen saturation (SpO2) <92% for more than 5 minutes.
  Regurgitation defined by visualized gastric contents requiring suctioning Aspiration defined by desaturation after regurgitation with suspicion of the anesthesiologist or CRNA that aspiration occurred.
Aspiration | Duration of Procedure
  Aspiration will be defined by desaturation (SpO2 <92) after regurgitation and inhalation of the gastric contents.
Duration of the endoscopic procedure | Duration of Procedure
  Insertion to removal of TEE probe
Sore throat | Duration of procedure up to 24 hours after the procedure ends.
  As described on a numerical rating scale, and at time 0, 2, and 24 hours 0= no sore throat , 1= mild sore throat, 2= moderate sore throat, 3= severe sore throat
Ease and comfort of advancing and operating the Endoscope by attending endoscopist | Duration of procedure
  The comfort of advancing and operating the endoscope rated by the attending endoscopist after the procedure via a 5 point Likert-type scale (0 = not at all satisfied, 1=slightly satisfied, 2=moderately satisfied, 3=very satisfied, 4 = completely satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Braunecker, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiew WA, Chen Q, Tan LZ. Use of LMAⓇ GastroTM in esophagogastroduodenoscopy and endoscopy. Korean J Anesthesiol. 2019 Dec;72(6):618-619. doi: 10.4097/kja.19163. Epub 2019 Jul 1. No abstract available. PMID 31257818
- [Background] Terblanche NCS, Middleton C, Choi-Lundberg DL, Skinner M. Efficacy of a new dual channel laryngeal mask airway, the LMA(R)Gastro Airway, for upper gastrointestinal endoscopy: a prospective observational study. Br J Anaesth. 2018 Feb;120(2):353-360. doi: 10.1016/j.bja.2017.11.075. Epub 2017 Dec 1. PMID 29406183
- [Background] Tran A, Thiruvenkatarajan V, Wahba M, Currie J, Rajbhoj A, van Wijk R, Teo E, Lorenzetti M, Ludbrook G. LMA(R) Gastro Airway for endoscopic retrograde cholangiopancreatography: a retrospective observational analysis. BMC Anesthesiol. 2020 May 13;20(1):113. doi: 10.1186/s12871-020-01019-5. PMID 32404136
- [Background] Schmutz A, Loeffler T, Schmidt A, Goebel U. LMA Gastro airway is feasible during upper gastrointestinal interventional endoscopic procedures in high risk patients: a single-center observational study. BMC Anesthesiol. 2020 Feb 8;20(1):40. doi: 10.1186/s12871-020-0938-9. PMID 32035477
- [Background] Hakim M, Bryant J, Miketic R, Williams K, Erdman SH, Shafy SZ, Kim SS, Tobias JD. Clinical Outcomes of a Modified Laryngeal Mask Airway (LMA(R) Gastro Airway) During Esophagogastroduodenoscopy in Children and Adolescents: A Randomized Study. Med Devices (Auckl). 2020 Sep 21;13:277-282. doi: 10.2147/MDER.S272557. eCollection 2020. PMID 33061677
- [Background] Waruingi D, Mung'ayi V, Gisore E, Wanyonyi S. A randomised controlled trial of the effect of laryngeal mask airway manometry on postoperative sore throat in spontaneously breathing adult patients presenting for surgery at a university teaching hospital. Afr Health Sci. 2019 Mar;19(1):1705-1715. doi: 10.4314/ahs.v19i1.47. PMID 31149001
- [Background] Seet E, Yousaf F, Gupta S, Subramanyam R, Wong DT, Chung F. Use of manometry for laryngeal mask airway reduces postoperative pharyngolaryngeal adverse events: a prospective, randomized trial. Anesthesiology. 2010 Mar;112(3):652-7. doi: 10.1097/ALN.0b013e3181cf4346. PMID 20179502
- [Background] Balmforth D, Smith A, Nagore D, Schilling R, O'Brien B. Can Transesophageal Echocardiography Be Performed Safely Using a Laryngeal Mask Airway During Atrial Fibrillation Ablation? J Cardiothorac Vasc Anesth. 2018 Apr;32(2):790-795. doi: 10.1053/j.jvca.2017.10.040. Epub 2017 Nov 2. PMID 29229253
- [Background] Salvi L, Pepi M. Pressure-assisted breathing through a laryngeal mask airway during transesophageal echocardiography. Anesth Analg. 1999 Dec;89(6):1591-2. doi: 10.1097/00000539-199912000-00070. No abstract available. PMID 10589667
- [Background] Ferson D, Thakar D, Swafford J, Sinha A, Sapire K, Arens J. Use of deep intravenous sedation with propofol and the laryngeal mask airway during transesophageal echocardiography. J Cardiothorac Vasc Anesth. 2003 Aug;17(4):443-6. doi: 10.1016/s1053-0770(03)00147-2. PMID 12968230
- [Background] Patrick Mayr N, Michel J, Wiesner G, Rumpf PM. Supraglottic airway device use for transoesophageal echocardiography during left atrial appendage occlusion. Anaesthesia. 2019 Mar;74(3):405-406. doi: 10.1111/anae.14597. No abstract available. PMID 30734949
- [Background] Saxena S, Aminian A, Nahrwold DA, Daper A. LMA Gastro Airway Seen Through the Eyes of a Cardiac Anesthesiologist. J Cardiothorac Vasc Anesth. 2019 Aug;33(8):2365-2366. doi: 10.1053/j.jvca.2019.04.014. Epub 2019 Apr 20. No abstract available. PMID 31101507
- See also: Power calculator for binary outcome non-inferiority trial. Sealed Envelope Ltd. 2012. Power calculator for binary outcome non-inferiority trial. [Online] [Accessed Sat Apr 03 2021]. — https://www.sealedenvelope.com/power/binary-noninferior/